CLINICAL TRIAL: NCT02915718
Title: A Randomized, Open, Controlled Clinical Study of Immunoadsorption Therapy for Dilated Cardiomyopathy
Brief Title: A Clinical Study of Immunoadsorption Therapy for Dilated Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiang Cheng, Professor, Chief Physician, Deputy Director, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XCheng
Record Dates: First submitted 2016-09-20; First posted 2016-09-27 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Dilated Cardiomyopathy
Keywords: dilated cardiomyopathy; immunoadsorption
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (Experimental): protein A immunoadsorption for 5 days
  Interventions: Procedure: protein A immunoadsorption
- control group (No Intervention): non intervention

INTERVENTIONS:
Procedure: protein A immunoadsorption — protein-A immunoadsorption for 5 days and i.v. IgG（0.5g/kg Body weight）substitution
  Other Names: plasma adsorption
  Arms: experimental group

SUMMARY:
Dilated cardiomyopathy (DCM) causes significant morbidity and mortality and is the third most common cause of heart failure and the most frequent reason for heart transplantation. The etiology of dilated cardiomyopathy(DCM) is complex. There is a growing body of literature suggesting that the humoral immune system activation and autoantibodies against myocardial generation play an important role in the progression of DCM. At present immunoadsorption technology has been successfully applied in autoimmune antibody removal treatment of a variety of diseases. And some applications of immunoadsorption(IA) in patients with DCM showed that immunoadsorption(IA) can indeed reduce the autoantibodies, improve symptoms and prognosis, but additional research is needed to identify indications and instruments for the IA treatment of DCM.

DETAILED DESCRIPTION:
40 patients randomly divided into 2 groups： experimental group and control group

experimental group：

Device: protein A immunoadsorption

protein-A immunoadsorption for 5 days and i.v.(intravenous injection) IgG(Immunoglobulin G）（0.5g/kg Body weight） substitution

control group：

non intervention

ELIGIBILITY:
Inclusion Criteria:

* Dilated cardiomyopathy
* LVEF <= 40% determined by contrast echocardiography
* NYHA(New York Heart Association) class II - IV
* Age 18-70
* Disease duration: symptomatic heart failure ≥ 6 months prior to screening date
* Treatment with Angiotensin-Converting Enzyme inhibitors(ACEI) or angiotensin II receptor blockers (ARB), beta-blockers, and aldosterone antagonists (the latter at the discretion of the attending physician), for at least 6 months and at stable doses for at least 2 months prior to screening date.
* β1 adrenergic receptor antibody positive
* The patient's informed consent

Exclusion Criteria:

* NYHA class IV patients who are bed-ridden and dependent upon parenteral medication
* Cardiac insufficiency resulting from another basic disease (e.g. coronary artery disease, ≥50% stenosis of major vessel as ascertained by coronary angiography performed more recent than three years before screening date, hypertensive heart disease, or valvular defects >second degree
* History of myocardial infarction
* Acute myocarditis according to Dallas criteria
* Endocrine disorder excluding insulin-dependent diabetes mellitus
* Implanted cardiac defibrillator (ICD) <1 month before screening date
* Cardiac resynchronization therapy (CRT) <6 months before screening date
* I.v. medication with inotropic drugs, vasodilators or repeated (>1/day) i.v. administration of diuretics.
* Active infectious disease, or signs of ongoing infection with C-reactive protein(CRP) >10mmol/L
* Impaired renal function (serum creatinine >220 µmol/L)
* Any disease requiring immunosuppressive drugs
* Anaemia (haemoglobin below 90 g/L) due to other causes than congestive heart failure(CHF)
* Pregnancy or lactation, or childbearing potential without appropriate contraception
* Alcohol or drug abuse
* Presence of a malignant tumour, or remission of malignancy < 5 years
* Refusal of the patient to provide consent
* Suspected poor capability to follow instructions and cooperate
* Another life-threatening disease with poor prognosis (survival less than 2 years)
* Participation in any other clinical study within less than 30 days prior to screening date
* Previous treatments with IA or immunoglobulin
* Contraindications for application of the echocardiography contrast agent used (in accordance to the product specification).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-10; Primary Completion 2022-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) at rest | six months
  determined by contrast echocardiography

SECONDARY OUTCOMES:
LVEF at rest | 1 year
  determined by contrast echocardiography
Reduction of brain natriuretic peptides (BNP) or N-terminal pro-Brain Natriuretic Peptide(NT pro-BNP) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tian Xie, master, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ameling S, Herda LR, Hammer E, Steil L, Teumer A, Trimpert C, Dorr M, Kroemer HK, Klingel K, Kandolf R, Volker U, Felix SB. Myocardial gene expression profiles and cardiodepressant autoantibodies predict response of patients with dilated cardiomyopathy to immunoadsorption therapy. Eur Heart J. 2013 Mar;34(9):666-75. doi: 10.1093/eurheartj/ehs330. Epub 2012 Oct 25. PMID 23100283
- [Background] Dandel M, Wallukat G, Englert A, Lehmkuhl HB, Knosalla C, Hetzer R. Long-term benefits of immunoadsorption in beta(1)-adrenoceptor autoantibody-positive transplant candidates with dilated cardiomyopathy. Eur J Heart Fail. 2012 Dec;14(12):1374-88. doi: 10.1093/eurjhf/hfs123. Epub 2012 Aug 14. PMID 22892122